CLINICAL TRIAL: NCT04722510
Title: Effect of Repeated Transcranial Magnetic Stimulation on Aggressive Impulsive Behavior in Patients With Borderline Personality Disorder in a Social Exclusion Paradigm.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI/C/088/2016
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect of repeated TMS on aggressive impulse behavior in patients with BPD. (Experimental): A protocol of 15 sessions of repeated Transcranial Magnetic Stimulation at 1 Hz on right dorsolateral prefrontal cortex.
  Interventions: Device: repeated transcranial magnetic stimulation

INTERVENTIONS:
Device: repeated transcranial magnetic stimulation — Transcranial magnetic stimulation is a non-invasive brain modulation technique that has proven to be a useful study and treatment tool in neuropsychiatric disorders. This technique allows to increase (with high frequency protocol, > 1 Hz) or decrease (with low frecuency protocols, 1 hz or less) neuronal excitability in a focused cortical area.

SUMMARY:
Patients with a main diagnosis of borderline personality disorder will be recruited and will be randomized for the application of low frequency repeated transcranial magnetic stimulation (rTMS) protol or sham rTMS protocol. A pre-treatment and post-treatment measurement of the severity of BPD symptoms, impulsivity, and aggressive behavior will be carried out in all participants using self-administered questionnaires. All participants will be asked to participate in a passing ball game (Cyberball) with the intention of investigating aspects related to social inclusion / exclusion and measurements will be made regarding planning using the maze test. Participation in the Cyberball and the assessment of the planning will be carried out before and after the application of the treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient consultant in the Instituto Nacional de Psiquiatría Ramón de la Fuente Muñiz.
* Main diagnosis of borderline personality disorder according to DSM-IV-TR.
* In the case of having some type of pharmacological treatment using SSRIs, antipsychotics and / or anticonvulsants, this should be maintained without modifications for at least 2 weeks prior to the start of the study and during the follow-up period.
* Comorbidity with some other personality disorder according to the SCID-II, with the exception of antisocial personality disorder.
* Acceptance of participation in the study by signing the informed consent.

Exclusion Criteria:

* Subjects who did not agree to participate.
* Diagnosis of current antisocial personality disorder, bipolar disorder, psychotic disorders, severe major depressive episode, substance use disorder (except nicotine), and post-traumatic stress disorder.
* Presence of any comorbid neurological disorder.
* Diagnosis of intellectual disability.
* Subjects in whom the use of rTMS is contraindicated: history of seizures, pregnancy, presence of pacemaker, heart disease, and presence of a metallic object.
* Electroencephalographic evidence of some type of abnormality in the excitability of the central nervous system (dysrhythmias, paroxysmal activity, graphical elements suggestive of epileptic activity, etc.).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-01-21 (Estimated); Study Completion 2021-01-21 (Estimated)

PRIMARY OUTCOMES:
Maneuver effect | 3 weeks
  To determine whether the application of a series of 15 sessions of low-frequency (1 Hz) repeated Transcranial Magnetic Stimulation applied to the right dorsolateral prefrontal cortex reduces the severity of impulse agressive behavior in subjects with BPD as measured by the impulsive / premeditated aggression scale.

CONTACTS AND LOCATIONS:
Overall Officials: JORGE GONZALEZ-OLVERA, PHD, Study Chair — Instituto Nacional de Psiquiatría Ramon de la Fuente Muñiz
Locations (1):
- Instituto Nacional de Psiquiatria Ramon de la Fuente Muñiz, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
In case of being requested